CLINICAL TRIAL: NCT06664658
Title: Assessment of the Impact of Two Different PEEP Levels on Pulmonary Functions in Laparoscopic Cholecystectomy Using Ultrasound
Brief Title: Lung Ultrasound, Cholecystectomy, Atelectasis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul Medeniyet University (Other)
Responsible Party: Principal Investigator, Ezgi POLAT, Principal Investigator, Istanbul Medeniyet University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IRB: Approval No. 2022/0257
Record Dates: First submitted 2024-10-18; First posted 2024-10-29 (Actual); Last update posted 2024-10-29 (Actual); Status verified 2024-10

CONDITIONS: Laparoscopic Cholecystectomy
Keywords: General Anesthesia, Lung Ultrasonography, PEEP, Pneumoperitoneum, Atelectasis
MeSH Terms: conditions — Pneumoperitoneum; Pulmonary Atelectasis

STUDY DESIGN:
Intervention Model Description: two groups:
  * PEEP 5 cm H2O
  * PEEP 10 cm H2O
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- PEEP 5 (Active Comparator): Patients are in the group undergoing PEEP 5 cm h2o during surgery
  Interventions: Procedure: peep 5
- peep 10 (Active Comparator): Patients are in the group undergoing PEEP 10 cm h2o during surgery
  Interventions: Procedure: peep 10

INTERVENTIONS:
Procedure: peep 5 — he patients included in the study were divided into 2 groups. Among the patients who were going to be operated, 5 PEEP were applied to Group I (n=30) cases, and 10 PEEP to Group II (n=30) cases during ventilation with anesthesia device. All patients were evaluated by transthoracic lung ultrasonography before anesthetic induction, after tracheal intubation, after pneumoperitoneum, and 15 minutes after recovery from anesthesia. According to the lung USG protocol, a total of 6 regions, including 2 quadrants of each hemi-thorax anterior wall, 2 right and left lateral walls, and 2 quadrants of the posterior wall, a total of 12 regions in each patient were scanned, and the images were evaluated. According to the modified lung USG scoring system, each region was scored between 0-3 consistent with the degree of atelectasis
  Arms: PEEP 5
Procedure: peep 10 — he patients included in the study were divided into 2 groups. Among the patients who were going to be operated, 5 PEEP were applied to Group I (n=30) cases, and 10 PEEP to Group II (n=30) cases during ventilation with anesthesia device. All patients were evaluated by transthoracic lung ultrasonography before anesthetic induction, after tracheal intubation, after pneumoperitoneum, and 15 minutes after recovery from anesthesia. According to the lung USG protocol, a total of 6 regions, including 2 quadrants of each hemi-thorax anterior wall, 2 right and left lateral walls, and 2 quadrants of the posterior wall, a total of 12 regions in each patient were scanned, and the images were evaluated. According to the modified lung USG scoring system, each region was scored between 0-3 consistent with the degree of atelectasis
  Arms: peep 10

SUMMARY:
Atelectasis is an important complication that can be seen during general anesthesia, especially in patients with lung problems and in patients having pneumoperitoneum. Application of PEEP during anesthesia may reduce the incidence of atelectasis.Lung ultrasonography is a tool that is easily accessible, can be applied at the bedside, is non-invasive, does not cause radiation exposure, and is increasingly used in daily practice in operating rooms. In this study, it was aimed to evaluate the occurrence of atelectasis by using lung ultrasound, and to investigate the effectiveness of ultrasound in determining the risk of developing atelectasis in patients ventilated with different PEEP values during general anesthesia. The study was conducted in 60 patients aged 18 and over, from ASA I-III groups, who were planned to undergo laparoscopic cholecystectomy surgery at the Istanbul Medeniyet University Göztepe Training and Research Hospital General Surgery Clinic, and their written and verbal informed consents were obtained. The patients included in the study were divided into 2 groups. Among the patients who were going to be operated, 5 PEEP were applied to Group I (n=30) cases, and 10 PEEP to Group II (n=30) cases during ventilation with anesthesia device. All patients were evaluated by transthoracic lung ultrasonography before anesthetic induction, after tracheal intubation, after pneumoperitoneum, and 15 minutes after recovery from anesthesia. According to the lung USG protocol, a total of 6 regions, including 2 quadrants of each hemi-thorax anterior wall, 2 right and left lateral walls, and 2 quadrants of the posterior wall, a total of 12 regions in each patient were scanned, and the images were evaluated. According to the modified lung USG scoring system, each region was scored between 0-3 consistent with the degree of atelectasis. The total score was calculated for each patient. Hemodynamic follow-up of the patients was performed. Anesthesia times, surgery times, and pneumoperitoneum times were recorded and compared.

ELIGIBILITY:
Inclusion Criteria:

* Patients are aged 18 and over, from ASA I-III groups, who were planned to undergo laparoscopic cholecystectomy surgery

Exclusion Criteria:

* Patients who do not give consent
* Patients who have previously undergone thoracic surgery
* Patients with a body mass index > 40 kg/m²
* Patients with severe COPD
* Patients with serious pulmonary diseases
* Patients diagnosed with obstructive sleep apnea syndrome
* ASA IV patients
* Patients with advanced cardiac and neurological diseases
* Patients with mental retardation and limited cooperation
* Patients who terminate their participation in the study for any reason during the trial
* Pediatric age group Pregnant women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2022-05-01 (Actual); Primary Completion 2022-08-31 (Actual); Study Completion 2022-09-15 (Actual)

PRIMARY OUTCOMES:
The study will terminate once a population of 60 patients is reached. | Postoperative 24 hours
  All patients were evaluated by transthoracic lung ultrasonography before anesthetic induction, after tracheal intubation, after pneumoperitoneum, and 15 minutes after recovery from anesthesia. According to the lung USG protocol, a total of 6 regions, including 2 quadrants of each hemi-thorax anterior wall, 2 right and left lateral walls, and 2 quadrants of the posterior wall, a total of 12 regions in each patient were scanned, and the images were evaluated. According to the modified lung USG scoring system, each region was scored between 0-3 consistent with the degree of atelectasis

CONTACTS AND LOCATIONS:
Locations (2):
- Turkey (Türkiye) (2):
  - Turkey Istanbul Medeniyet University Faculty of Medicine Department of Anesthesiology and Reanimation, Istanbul, Kadikoy
  - Istanbul Medeniyet Universty, Istanbul, kadıköy

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Yu X, Zhai Z, Zhao Y, Zhu Z, Tong J, Yan J, Ouyang W. Performance of Lung Ultrasound in Detecting Peri-Operative Atelectasis after General Anesthesia. Ultrasound Med Biol. 2016 Dec;42(12):2775-2784. doi: 10.1016/j.ultrasmedbio.2016.06.010. Epub 2016 Sep 14. PMID 27639431